CLINICAL TRIAL: NCT05797675
Title: Osseodensification Plus Platelet Rich Fibrin With Simultaneous Implant Installation in Closed Sinus Lift : A Randomized Control Trial.
Brief Title: Osseodensification Plus Platelet Rich Fibrin With Simultaneous Implant Installation in Closed Sinus Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, hadeel bassam albahar, dr, Arab American University (Palestine)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAUP
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Oral Sinus
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Implant therapy and closed sinus lifting with A-PRF
  Interventions: Procedure: prf + osseodensification

INTERVENTIONS:
Procedure: prf + osseodensification — prf+ osseodensification in close sinus lift
  Other Names: platelet concentrates,

SUMMARY:
12 patients with indirect sinus lift will be selected with RBH>5mm , surgical procedure

=osseodensification + Prf+ implant .

1. versah drilling system (osseodensefication technique )will be used , moreover Prf will be prepared by Blood collected in PRF tubes from patients then centrifuge (1300rpm ,14min ) .
2. primary stability will be measured using Resonance Frequency Analysis by Osstellimmediately and after 6 Mn .
3. CBCT will be taken before surgery , perioapical x-ray immediately after surgery and CBCT at 6m follow up to be apple to see the differences regarding bone quality and volume.

ELIGIBILITY:
Inclusion Criteria:

- medically fit non pregnant no sinus pathology

Exclusion Criteria:

* young patients under 18
* sinus pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
secondary stability of implant | 6 months
  by osstel
bone density | 6 months
  measuring and evaluating bone density by cbct

CONTACTS AND LOCATIONS:
Overall Officials: hadeel albahar, master, Principal Investigator — Arab American University
Locations (1):
- Hadeel Albahar, Nablus, Palestinian Territories